CLINICAL TRIAL: NCT04573361
Title: Access to Chiropractic Care During the State of Emergency Generated by the COVID-19 Pandemic in Spain: a Pragmatic Controlled Trial
Brief Title: Access to Chiropractic Care During the COVID-19 Healthcare Emergency in Spain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Centro Universitario Maria Cristina (Other)
Collaborators: Université du Québec à Trois-Rivières (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiroCOVID19
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Musculoskeletal Pain; Disability Physical; Psychological Distress
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Three arms depending on the access to chiropractic care (no access, one visit or more than one) during the 14-days period of the trial. Measures were taken at the beginning and at the end of the 14-day period.
Masking Description: Care was provided by chiropractors,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Control (No Intervention): Patients having no access to chiropractic treatment during the trial
- Group Chiropractic Care one session (Experimental): Patients having access to in-person chiropractic treatment once during the trial
  Interventions: Other: Chiropractic care (one visit)
- Group Chiropractic Care multiple sessions (Experimental): Patients having access to in-person chiropractic treatment more than once during the trial
  Interventions: Other: Chiropractic care (more than one visit)

INTERVENTIONS:
Other: Chiropractic care (one visit) — One visit to the chiropractor based on the use of spinal manipulative therapy, mobilization and other forms of manual therapy, exercise therapy, patient education, advice and reassurance
  Other Names: Chiropractic Tx1
  Arms: Group Chiropractic Care one session
Other: Chiropractic care (more than one visit) — More than one visit to the chiropractor based on the use of spinal manipulative therapy, mobilization and other forms of manual therapy, exercise therapy, patient education, advice and reassurance
  Other Names: Chiropractic Tx2
  Arms: Group Chiropractic Care multiple sessions

SUMMARY:
This is a pragmatic controlled clinical trial taking place in the first phase of COVID-19 lockdown re-opening in Spain. Patients of 52 chiropractic clinics were invited to participate in a pseudo-random order (one out of every three contacted patients) as they were contacted to either schedule an appointment with their current chiropractor or not, depending on the clinic's and the patient's availability. Patients would receive chiropractic in-person care (one or more than one visits) or no care at all, for a two-week period. According to the care received, they were assigned to one of three groups (receiving no care, receiving care once, and more than once). Participants filled an online questionnaire with self-reported outcome-measures at the beginning of the two week period. A follow-up questionnaire was completed 14 days after.

ELIGIBILITY:
Inclusion Criteria:

* chiropractic patients active when lockdown was declared, over the age of 14

Exclusion Criteria:

* new patients in the clinic, patients with no current pain at the time of the trial

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 723 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 14 days
  Numerical rating scale (0-10, 0 meaning no pain, 10 meaning worst pain imaginable)
Pain frequency | 14 days
  Likert Scale from better (1) to worst (4) outcomes, 1: occasionally, 4: constantly
Pain evolution | 14 days
  Likert Scale of self-perceived improvement, from better (1) to worst (5) outcomes, 1: much better, 5: much worse
Pain interference | 14 days
  Validated subscale form the Brief Pain Inventory, 6 categories from 0 to 10 each, the lower, the better outcomes, out of a minimal of 0 and total of 60.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | 14 days
  Validated questionnaire. Short version 4 items, Likert scale from 0 to 4, lowest score (0) better outcomes, highest score (16) worst outcomes
Tampa Scale Kinesiophobia | 14 days
  Validated questionnaire. Short version 11 items, Likert scale from 1 to 4, lowest score (11) better outcomes, highest score (44) worst outcomes
General Anxiety Disorder scale | 14 days
  Validated questionnaire 7 items, Likert scale from 0 to 3, lowest score (0) better outcomes, highest score (21) worst outcomes
Intolerance of Uncertainty Scale | 14 days
  Validated questionnaire. Short version 12 items, Likert scale from 1 to 5, lowest score (12) better outcomes, highest score (60) worst outcomes
General Self-Efficacy scale | 14 days
  Validated questionnaire 10 items, Likert scale from 1 to 10, lowest score (10) WORST outcomes, highest score (100) BETTER outcomes
Fear of Illness and Virus Evaluation | 14 days
  Questionnaire, subscale 10 items, Likert scale from 1 to 4, lowest score (1) WORST outcomes, highest score (40) BETTER outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Arantxa Ortega de Mues, PhD, Principal Investigator — Madrid College of Chiropractic - Real Centro Universitario Maria Cristina
Locations (1):
- Real Centro Universitario María Cristina, El Escorial, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
All collected IPD will be shared, though a next phase of the study is being debated, which is why we are still undecided.